CLINICAL TRIAL: NCT04833738
Title: Subakromiyal sıkışma Sendromunda Hyaluronik Asit, Kortikosteroid ve Elektroterapi
Brief Title: Hyaluronic Acid, Corticosteroid and Electrotherapy in Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şeyhmus KAPLAN (Other)
Responsible Party: Sponsor-Investigator, Şeyhmus KAPLAN, Department of Sports Medicine, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yuzuncu Yil University
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Subacromial Impingement; Pain, Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Hyaluronic Acid; Triamcinolone; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electrotherapy (Active Comparator)
  Interventions: Other: Electrotherapy
- corticosteroid (Active Comparator)
  Interventions: Drug: Corticosteroids Triamcinolone Acetonide
- hyaluronic acid (Active Comparator)
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Hyaluronic acid
  Arms: hyaluronic acid
Drug: Corticosteroids Triamcinolone Acetonide — triamcinolone acetonide, 40 mg/ml, single dose
  Arms: corticosteroid
Other: Electrotherapy — electrotherapy
  Arms: Electrotherapy

SUMMARY:
Background: Electrotherapy, corticosteroid, and hyaluronic acid have been used to treat subacromial impingement syndrome. However, we need to compare treatment options to provide the optimal results. This study aims to compare the effect of hyaluronic acid, corticosteroid, and electrotherapy in subacromial impingement syndrome.

Design: Ninety five patients were randomised into three equal groups according to treatment types. Hyaluronic acid (20 mg/2ml, three times one week apart) or corticosteroid (triamcinolone acetonide, 40 mg/ml, single dose) treatments were applied as subacromial injections. Electrotherapy consisted of 14 sessions TENS (20 min.), hotpack (20 min.) and ultrasound (1.5watt/cm2, 1 MHz, 6 min.). Patients were evaluated before treatment, one and four weeks post end of treatment. Visual Analogue Scale (VAS), range of motion (ROM), and Shoulder Disability Questionnaire (SDQ) were used as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of subacromial impingement syndrome

Exclusion Criteria:

* Patients aged <20 or >50 years or who have the following medical conditions were excluded: physical therapy or injection in the past 6 months, shoulder instability, acute trauma, adhesive capsulitis, psychiatric illness, diabetes mellitus, malignancy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2014-05-28 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 min.
  Higher scores represent higher level of shoulder pain.
range of motion | 5 min.
  Higher scores represent lower level of shoulder function.
Shoulder Disability Questionnaire | 15 min
  Higher scores represent higher level of shoulder pain.

IPD SHARING:
Plan to Share IPD: No